CLINICAL TRIAL: NCT04619654
Title: Visual Acuity, Refractive Predictability, and Patient Reported Quality of Vision in Subjects Implanted With a Trifocal IOL With Stable Mild Open-Angle Glaucoma Undergoing Concurrent Minimally Invasive Glaucoma Surgery
Brief Title: Visual Outcomes With a Trifocal IOL in Subjects With Open-angle Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vold Vision P.L.L.C (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PanOptix Trifocal 001, Rev A
Record Dates: First submitted 2020-11-02; First posted 2020-11-06 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-05

CONDITIONS: Cataract; IOL; Glaucoma, Open-Angle
Keywords: PanOptix; Trifocal IOL; Glaucoma; MIGS
MeSH Terms: conditions — Cataract; Glaucoma, Open-Angle; Glaucoma | interventions — Cataract Extraction

STUDY DESIGN:
Intervention Model Description: Prospective single arm open label descriptive case series
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Cataract Surgery with concurrent MIGS (Experimental)
  Interventions: Procedure: Cataract surgery with implantation of trifocal IOL combined with trabecular scaffold

INTERVENTIONS:
Procedure: Cataract surgery with implantation of trifocal IOL combined with trabecular scaffold — Cataract surgery with implantation of the PanOptix IOL combined with minimally invasive glaucoma surgery utilizing the Hydrus Microstent

SUMMARY:
This study will examine the visual outcomes of subjects undergoing cataract surgery and minimally invasive glaucoma surgery with the implantation of a trifocal intraocular lens.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects 45 years of age or older
2. A visually significant cataract
3. Diagnosis of mild OAG

   * Vertical C/D ratio of less than or equal to 0.8
   * VF characteristics consistent with glaucoma with mean deviation not worse than -6.00 dB and without fixation threatening scotoma AND/OR with nerve abnormalities consistent with glaucoma (rim notching, rim thinning, disc hemorrhage, nerve fiber layer loss)
   * Medicated IOP 25 of less than or equal to mmHg on 1-3 medications
   * If treatment naïve (before glaucoma treatment) IOP between 21 and 35 mmHg
4. Glaucoma must be judged as stable by investigator based on review of subject medical records

   * Stable VF at least 1 year prior to surgery
   * Stable nerve fiber layer at least 1 year prior to surgery
   * IOP stable on current medication regimen at least 3 months prior to surgery
5. Shaffer grade of greater than III in all quadrants
6. Potential of good best corrected visual acuity at distance in the investigator's judgement of at least 0.1 logMAR (20/25) postoperatively
7. Able and willing to comply with follow up visits
8. Understands and signs the informed consent

Exclusion Criteria:

1. Previous incisional glaucoma surgery or cilio-ablative surgery
2. Prior laser trabeculoplasty within 90 days of surgery
3. Pseudoexfoliative, angle closure, uveitic, congenital, traumatic, angle recession, or neovascular glaucoma.
4. Moderate glaucoma with VF mean deviation between -6.00 dB and -12.00 dB
5. Severe and/or progressive glaucoma defined as

   * VF mean deviation worse than -12.00 dB
   * Consistent worsening of visual field on review of subject medical records
   * Consistent and progressive thinning of nerve fiber layer on review of subject medical records
   * Uncontrolled IOP on maximum glaucoma medications
   * Historically poor IOP control with medical therapy
   * Severe focal notching of the optic nerve rim
   * Expectation for future need of incisional glaucoma surgery
6. Ocular pathology or other medical condition which, in the investigator's judgment places the subject at increased risk of complications or significant vision loss during study period.
7. Ocular pathology that in the investigator's judgment may impact visual acuity postoperatively, i.e. significant ocular surface disease, corneal scarring, blepharitis, epiretinal membrane, macular degeneration, history of significant ocular trauma with sequela, etc.
8. Pregnant or breastfeeding women
9. Prior refractive surgery e.g. LASIK, RK, PRK, etc.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Mean Photopic Monocular Best Corrected Distance Visual Acuity (DCVA) (4 meters) logMAR | 3 months

SECONDARY OUTCOMES:
Mean Photopic Monocular Best Distance Corrected Intermediate Visual Acuity (DCIVA) (60 cm) logMAR | 3 months
Mean Photopic Monocular Best Distance Corrected Near Visual Acuity (DCNVA) (40 cm) logMAR | 3 months
Mean Photopic Monocular Uncorrected Distance Visual Acuity (UCDVA) (4 meters) logMAR | 3 months
Mean Photopic Monocular Uncorrected Intermediate Visual Acuity (UCIVA) (60 cm) logMAR | 3 months
Mean Photopic Monocular Uncorrected Near Visual Acuity (UCNVA) (40 cm) logMAR | 3 months
Mean Photopic Binocular Best Corrected Distance Visual Acuity (DCVA) (4 meters) logMAR | 3 months
Mean Photopic Binocular Best Distance Corrected Intermediate Visual Acuity (DCIVA) (60 cm) logMAR | 3 months
Mean Photopic Binocular Best Distance Corrected Near Visual Acuity (DCNVA) (40 cm) logMAR | 3 months
Mean Photopic Binocular Uncorrected Distance Visual Acuity (UCDVA) (4 meters) logMAR | 3 months
Mean Photopic Binocular Uncorrected Intermediate Visual Acuity (UCIVA) (60 cm) logMAR | 3 months
Mean Photopic Binocular Uncorrected Near Visual Acuity (UCNVA) (40 cm) logMAR | 3 months
Mean Photopic Binocular Best Corrected Distance Low Contrast Visual Acuity (25%) (4 meters) logMar | 3 months
Mean Mesopic Binocular Best Corrected Distance Low Contrast Visual Acuity (25%) (4 meters) logMar | 3 months

OTHER OUTCOMES:
Mean Postoperative Refractive Spherical Equivalent | 3 months
Absolute Prediction Error | 3 months
  Difference from postoperative refraction from preoperative biometry
Quality of Vision Questionnaire (QoV) | 3 months
  Grading of dysphotopsia
Spectacle-Dependence questionnaire | 3 months
  Gauging spectacle independence postoperatively
Mean preoperative IOP versus postoperative IOP | 3 months
Glaucoma Mean preoperative medications versus postoperative medications | 3 months
Percentage of patients with an IOP of less than or equal to18 mmHg and less than or equal to15 mm Hg on no glaucoma medications postoperatively | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Vold Vision P.L.L.C., Fayetteville, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No
Plan to publish results in open access peer reviewed journal